CLINICAL TRIAL: NCT04428697
Title: Sungurtekin Technique vs. Closed Lateral Internal Sphincterotomy for Chronic Fissure-in-Ano: A Prospective, Randomized, Controlled Trial of a New Technique
Brief Title: Sungurtekin Technique vs. Closed Lateral Internal Sphincterotomy Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Hulya Sungurtekin, Professor in Anesthesiology and Critical Care, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Sungurtekin 01
Record Dates: First submitted 2020-05-22; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Anal Fissure
Keywords: Fissure-in-ano; Sphincterotomy; İncontinence; Surgical technique
MeSH Terms: conditions — Fissure in Ano

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessor doesn't know the type of the surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sungurtekin Technique (Experimental): Sungurtekin technique was performed through the base of the posterior fissure; thus, no additional incision was necessary in the lithotomy position. The mucosa was dissected along the submucosal plane, starting at the hypertrophic papilla, and extended for 1.5 cm. After identifying both the internal and external sphincters completely, under direct vision, a 0.5-cm section of the bottom part of the internal anal sphincter was measured and marked with a ruler. This section was preserved during the operation in a standard fashion for all patients . Next, the internal sphincter bundle was measured with a sterile scale and a mark was placed at 1 cm towards the proximal end. The internal sphincter bundle was elevated with a right angle clamp, then cut with cautery . The operation was completed with meticulous hemostasis and additional suturing (3/0 absorbable suture) of the proximally dissected mucosal flap underlying the muscularis layer
  Interventions: Procedure: Sungurtekin Technique
- Closed Lateral Internal Sphincterotomy (Active Comparator): The sphincterotomy was performed through a new incision, guided by the surgeon's finger, as described by Boulos et al Boulos PB, Araujo JG. Adequate internal sphincterotomy for chronic anal fissure: subcutaneous or open technique? The British journal of surgery 1984;71:360-2.
  Interventions: Procedure: Sungurtekin Technique

INTERVENTIONS:
Procedure: Sungurtekin Technique — Sungurtekin technique was performed through the base of the posterior fissure; thus, no additional incision was necessary in the lithotomy position. The mucosa was dissected along the submucosal plane, starting at the hypertrophic papilla, and extended for 1.5 cm, a 0.5-cm section of the bottom part of the internal anal sphincter was measured and marked with a ruler. Next, the internal sphincter bundle was measured with a sterile scale and a mark was placed at 1 cm towards the proximal end. The internal sphincter cut with cautery .

SUMMARY:
BACKGROUND: Currently, the lateral internal sphincterotomy is the treatment of choice for a chronic anal fissure. However, the length of the internal sphincter incision varies, due to lack of standardization. Insufficient length increases the risk of recurrence.

OBJECTIVE: To compare a new ultra-modified internal sphincterotomy technique to the closed lateral sphincterotomy for treating chronic anal fissures, based on internal anal sphincter function and postoperative complications.

DESIGN: Prospective, randomized, controlled trial (block randomization method) SETTING: Pamukkale University hospital in Denizli-Turkey PARTICIPANTS: 200 patients with chronic anal fissures INTERVENTION: Patients were randomly assigned to receive either Sungurtekin technique (n = 100; ultra-modified group), or the closed lateral internal sphincterotomy (n = 100; closed-lateral group). Follow-up was 2 years.

MAIN OUTCOME MEASURES: The primary outcome was chronic anal fissure healing. The secondary outcomes were complications, visual analog scale pain scores, sphincter pressures, and incontinence scores.

DETAILED DESCRIPTION:
Although the lateral internal sphincterotomy is the treatment of choice for CAF, it has several drawbacks. First, the lower portion of the internal sphincter is nested in the lowermost part of the anus. Thus, an incision from the fissure base up to the dentate line removes support to the inner sphincter structure on the incision site. In our opinion; this is the main cause of different levels of incontinence developing in the postoperative period. Second, the internal sphincter muscle is shorter in women than in men. Therefore, women are at higher risk of postoperative anal incontinence than men. Third, because the lateral internal sphincterotomy is not standardized, the length of the internal sphincter incision varies, depending on the surgeon's discretion and competency. Fourth, an incision that is too short increases in the risk of recurrence.

The investigators believe that this observation could be explained by the fact that the length of the incision required for a lateral internal sphincterotomy procedure has not been standardized

ELIGIBILITY:
Inclusion Criteria:

Patients with CAFs that had failed conservative therapy and required surgical treatment

-

Exclusion Criteria:

* Patients who have a low resting anal pressure in manometric study (lower than 40 mmHg)
* Recurrent anal fissure
* Fissure location other than the posterior anal canal
* Fissure due to inflammatory bowel or infectious disease
* Acute anal fissure,
* Fissure due to chronic diarrhea or anal stenosis
* Anorectal malignancy
* Patients undergone pelvic radiotherapy
* Pregnancy
* Patients with history of diabetes, neurological disease and spinal cord lesions
* Previous episiotomy history
* Painless fissures

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 1-24 month
  It has been reported in the literature that healing was completed in 6-8 weeks in patients undergoing this operation. During this period, it was accepted that the fissure was no longer detected as a visual examination finding and that patient complaints disappeared.
Postoperatif pain | Postopetaive 3th day
  The patients asked to record postoperative pain scores with VAS(Visual Analog Scale)Graded from 0.0 to 10.0. and measured postoperative day 3 .As low as possible this pain score value indicates that the patient is exposed to less pain.
Incontinence Rate | 12th month
  Pre and postoperative fecal continence were scored using the Cleveland Clinic Florida Fecal Incontinence (CCF-FI) scores. Cleveland Clinic Florida (CCF) scores were used to assess the severity of fecal incontinence at baseline, and at 12 months. The scores from 0 indicate perfect continence to a maximum of 20 indicates complete incontinence The CCF FI scale combines loss of flatus, liquid and solid stool, use of a pad and the impact on the quality of life a assess the severity of fecal incontinence.
Complications | 1-24 month
  Urinary retansion,ecchymosis,itching,bleeding,abscess,fistula has been accepted as postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Ugur Sungurtekin, MD, Study Director — Pamukkale University Department Of Surgery,Colorectal Surgery Division

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tocchi A, Mazzoni G, Miccini M, Cassini D, Bettelli E, Brozzetti S. Total lateral sphincterotomy for anal fissure. Int J Colorectal Dis. 2004 May;19(3):245-9. doi: 10.1007/s00384-003-0525-9. Epub 2003 Sep 9. PMID 13680282
- [Result] Gandomkar H, Zeinoddini A, Heidari R, Amoli HA. Partial lateral internal sphincterotomy versus combined botulinum toxin A injection and topical diltiazem in the treatment of chronic anal fissure: a randomized clinical trial. Dis Colon Rectum. 2015 Feb;58(2):228-34. doi: 10.1097/DCR.0000000000000307. PMID 25585082
- [Result] Salih AM. Chronic anal fissures: Open lateral internal sphincterotomy result; a case series study. Ann Med Surg (Lond). 2017 Feb 14;15:56-58. doi: 10.1016/j.amsu.2017.02.005. eCollection 2017 Mar. PMID 28239456
- [Result] Liang J, Church JM. Lateral internal sphincterotomy for surgically recurrent chronic anal fissure. Am J Surg. 2015 Oct;210(4):715-9. doi: 10.1016/j.amjsurg.2015.05.005. Epub 2015 Jun 27. PMID 26231724
- [Result] Wiley M, Day P, Rieger N, Stephens J, Moore J. Open vs. closed lateral internal sphincterotomy for idiopathic fissure-in-ano: a prospective, randomized, controlled trial. Dis Colon Rectum. 2004 Jun;47(6):847-52. doi: 10.1007/s10350-004-0530-2. Epub 2004 May 6. PMID 15129311
- [Result] Gupta V, Rodrigues G, Prabhu R, Ravi C. Open versus closed lateral internal anal sphincterotomy in the management of chronic anal fissures: a prospective randomized study. Asian J Surg. 2014 Oct;37(4):178-83. doi: 10.1016/j.asjsur.2014.01.009. Epub 2014 Mar 14. PMID 24637183
- [Result] Alawady M, Emile SH, Abdelnaby M, Elbanna H, Farid M. Posterolateral versus lateral internal anal sphincterotomy in the treatment of chronic anal fissure: a randomized controlled trial. Int J Colorectal Dis. 2018 Oct;33(10):1461-1467. doi: 10.1007/s00384-018-3087-6. Epub 2018 May 19. PMID 29779044
- [Result] Mentes BB, Guner MK, Leventoglu S, Akyurek N. Fine-tuning of the extent of lateral internal sphincterotomy: spasm-controlled vs. up to the fissure apex. Dis Colon Rectum. 2008 Jan;51(1):128-33. doi: 10.1007/s10350-007-9121-3. Epub 2007 Dec 18. PMID 18085337
- [Result] Murad-Regadas SM, Fernandes GO, Regadas FS, Rodrigues LV, Pereira Jde J, Regadas Filho FS, Dealcanfreitas ID, Holanda Ede C. How much of the internal sphincter may be divided during lateral sphincterotomy for chronic anal fissure in women? Morphologic and functional evaluation after sphincterotomy. Dis Colon Rectum. 2013 May;56(5):645-51. doi: 10.1097/DCR.0b013e31827a7416. PMID 23575405
- [Result] Tsunoda A, Takahashi T, Kusanagi H. Fissurectomy with vertical non-full-thickness sphincterotomy for chronic anal fissure. Tech Coloproctol. 2019 Oct;23(10):1009-1013. doi: 10.1007/s10151-019-02087-7. Epub 2019 Sep 24. No abstract available. PMID 31552509
- [Result] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Result] Boulos PB, Araujo JG. Adequate internal sphincterotomy for chronic anal fissure: subcutaneous or open technique? Br J Surg. 1984 May;71(5):360-2. doi: 10.1002/bjs.1800710517. PMID 6722464
- [Result] Stewart DB Sr, Gaertner W, Glasgow S, Migaly J, Feingold D, Steele SR. Clinical Practice Guideline for the Management of Anal Fissures. Dis Colon Rectum. 2017 Jan;60(1):7-14. doi: 10.1097/DCR.0000000000000735. No abstract available. PMID 27926552
- [Result] Cross KL, Massey EJ, Fowler AL, Monson JR; ACPGBI. The management of anal fissure: ACPGBI position statement. Colorectal Dis. 2008 Nov;10 Suppl 3:1-7. doi: 10.1111/j.1463-1318.2008.01681.x. No abstract available. PMID 18954306
- [Result] Brady JT, Althans AR, Neupane R, Dosokey EMG, Jabir MA, Reynolds HL, Steele SR, Stein SL. Treatment for anal fissure: Is there a safe option? Am J Surg. 2017 Oct;214(4):623-628. doi: 10.1016/j.amjsurg.2017.06.004. Epub 2017 Jul 5. PMID 28701263
- [Result] Manoharan R, Jacob T, Benjamin S, Kirishnan S. Lateral Anal Sphincterotomy for Chronic Anal Fissures- A Comparison of Outcomes and Complications under Local Anaesthesia Versus Spinal Anaesthesia. J Clin Diagn Res. 2017 Jan;11(1):PC08-PC12. doi: 10.7860/JCDR/2017/21779.9299. Epub 2017 Jan 1. PMID 28274000
- [Result] Garcia-Granero E, Sanahuja A, Garcia-Botello SA, Faiz O, Esclapez P, Espi A, Flor B, Minguez M, Lledo S. The ideal lateral internal sphincterotomy: clinical and endosonographic evaluation following open and closed internal anal sphincterotomy. Colorectal Dis. 2009 Jun;11(5):502-7. doi: 10.1111/j.1463-1318.2008.01645.x. Epub 2008 Jul 15. PMID 18637925
- [Result] Garcia-Granero E, Sanahuja A, Garcia-Armengol J, Jimenez E, Esclapez P, Minguez M, Espi A, Lopez F, Lledo S. Anal endosonographic evaluation after closed lateral subcutaneous sphincterotomy. Dis Colon Rectum. 1998 May;41(5):598-601. doi: 10.1007/BF02235266. PMID 9593242
- [Result] Lindsey I, Jones OM, Smilgin-Humphreys MM, Cunningham C, Mortensen NJ. Patterns of fecal incontinence after anal surgery. Dis Colon Rectum. 2004 Oct;47(10):1643-9. doi: 10.1007/s10350-004-0651-7. PMID 15540293
- [Result] Elsebae MM. A study of fecal incontinence in patients with chronic anal fissure: prospective, randomized, controlled trial of the extent of internal anal sphincter division during lateral sphincterotomy. World J Surg. 2007 Oct;31(10):2052-7. doi: 10.1007/s00268-007-9177-1. PMID 17665247
- [Result] Ribas Y, Hotouras A, Munoz-Duyos A, Murphy J, Chan CL. Sphincterotomy in women with chronic anal fissure? Are we asking for trouble? Dis Colon Rectum. 2014 Sep;57(9):e404. doi: 10.1097/DCR.0000000000000184. No abstract available. PMID 25101617
- [Result] Garg P, Garg M, Menon GR. Long-term continence disturbance after lateral internal sphincterotomy for chronic anal fissure: a systematic review and meta-analysis. Colorectal Dis. 2013 Mar;15(3):e104-17. doi: 10.1111/codi.12108. PMID 23320551
- [Result] Davies I, Dafydd L, Davies L, Beynon J. Long term outcomes after lateral anal sphincterotomy for anal fissure: a retrospective cohort study. Surg Today. 2014 Jun;44(6):1032-9. doi: 10.1007/s00595-013-0785-0. Epub 2013 Nov 19. PMID 24241581
- [Result] Ghayas N, Younus SM, Mirani AJ, Ghayasuddin M, Qazi A, Suchdev SD, Bakshi SK. FREQUENCY OF POST-OPERATIVE FAECAL INCONTINENCE IN PATIENTS WITH CLOSED AND OPEN INTERNAL ANAL SPHINCTEROTOMY. J Ayub Med Coll Abbottabad. 2015 Oct-Dec;27(4):878-82. PMID 27004344
- [Result] Casillas S, Hull TL, Zutshi M, Trzcinski R, Bast JF, Xu M. Incontinence after a lateral internal sphincterotomy: are we underestimating it? Dis Colon Rectum. 2005 Jun;48(6):1193-9. doi: 10.1007/s10350-004-0914-3. PMID 15906136